CLINICAL TRIAL: NCT03275493
Title: Chimeric Antigen Receptor T Cells Against CD19 With Cytokine Release Syndrome (CRS) Suppression Technology for Refractory/Relapsed CD19+ Acute Lymphoblastic Leukemia
Brief Title: CD19 CAR-T Cells With CRS Suppression Technology for r/r CD19+ Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UnicarTherapy201701
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-11

CONDITIONS: Acute Lymphoblastic Leukemia; CD19 Positive; Relapse; Refractory
Keywords: CD19+ ,CAR-T, CRS
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Cohort 1 (Experimental): This cohort will determine the safety and efficacy of CD19 CAR-T cells for CD19+ acute lymphoblastic leukemia
  Interventions: Biological: CD19 CAR-T cells
- Experimental: Cohort 2 (Experimental): This cohort will determine the safety and efficacy of CD19 CAR-T cells with CRS suppression technology for CD19+ acute lymphoblastic leukemia.
  Interventions: Biological: CD19 CAR-T cells with CRS suppression technology

INTERVENTIONS:
Biological: CD19 CAR-T cells — Express a Second Generation 4-1BB: CD19 CAR-T cells
  Arms: Experimental: Cohort 1
Biological: CD19 CAR-T cells with CRS suppression technology — Express a Second Generation 4-1BB:CD19 CAR-T cells with CRS suppression technology
  Arms: Experimental: Cohort 2

SUMMARY:
This is a single center,randomized ,two-cohorts, open-label ,phase 1/2 study to evaluate the efficacy and safety of T cells expressing CD19 chimeric antigen receptors treatment for relapsed/refractory CD19+ acute lymphoblastic leukemia patients.

DETAILED DESCRIPTION:
Relapsed/refractory CD19 + acute lymphoblastic leukemia patients were randomly enrolled in this study to compare the efficacy and safety between two cohorts: 1. CD19 CAR-T cells； 2. CD19 CAR-T cells with CRS suppression technology.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 to 65
2. Voluntary informed consent is given
3. Expected survival ≥12 weeks
4. Relapsed or refractory CD19+ acute leukemia, ineligible for allo-HSCT,or relapse after auto-HSCT
5. Organ function: (1)Left ventricular ejection fractions≥ 0.6 by echocardiography (2)ALT ≤3 times of ULN, or bilirubin <2.0 mg/dl (3)Creatinine < 2 mg/dl and less than 2.5 × normal for age (4)Prothrombin time and activated partial thromboplastin time < 2 times of ULN (5)Arterial oxygen saturation> 92%
6. Karnofsky score ≥ 60 ;
7. No history of combined chemotherapy in the recent 1 month and no immunotherapy in the recent 3 months;

Exclusion Criteria:

1. Uncontrolled active infections
2. Active hepatitis B or hepatitis C infection
3. HIV infection
4. History of myocardio infarction in the past 6 months, or history of severe arrhythmia
5. Congenital immunodeficiency
6. Pregnant or lactating women
7. History or presence of clinically relevant CNS pathology such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
8. Previous treatment with any gene therapy products

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe CRS | 30 days after infusion of CD19 CAR-T cells
  The safety of the CD19 CAR-T cells treatment will be evaluated and the maximum tolerated dose will be determined

SECONDARY OUTCOMES:
Overall response of CD19 CAR-T cells treatment who achieve morphology complete remission(CR) and MRD negativity. | 30 days after infusion of CD19 CAR-T cells
  The efficacy of the CD19 CAR-T cells infusion will be estimated based on the number of participants who have morphology complete remission(CR) and MRD negativity following the CD19 CAR- T cells infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The first affiliated hospital of soochow university, Suzhou, Jiangsu, China

REFERENCES:
- [Derived] Gong WJ, Qiu Y, Li MH, Chen LY, Li YY, Yu JQ, Kang LQ, Sun AN, Wu DP, Yu L, Xue SL. Investigation of the risk factors to predict cytokine release syndrome in relapsed or refractory B-cell acute lymphoblastic leukemia patients receiving IL-6 knocking down anti-CD19 chimeric antigen receptor T-cell therapy. Front Immunol. 2022 Aug 29;13:922212. doi: 10.3389/fimmu.2022.922212. eCollection 2022. PMID 36105799
- [Derived] Hua J, Zhang J, Zhang X, Wu X, Zhou L, Bao X, Han Y, Miao M, Li C, Fu C, Chen S, Tang X, Wu D, Qiu H. Donor-derived anti-CD19 CAR T cells compared with donor lymphocyte infusion for recurrent B-ALL after allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2021 May;56(5):1056-1064. doi: 10.1038/s41409-020-01140-6. Epub 2020 Nov 24. PMID 33235353